CLINICAL TRIAL: NCT06063798
Title: Comparison of Flow-Controlled Ventilation With EVONE Tritube and High Frequency Jet Ventilation in Patients Undergoing Laryngotracheal Surgery
Brief Title: Respiratory Effects of Flow-Controlled Ventilation and Jet Ventilation in Patients Undergoing Laryngotracheal Surgery
Acronym: Flowjet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Dr. Gergely Albu, Principal investigator, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BASEC2022-D0078; SNCTP000005183 (Registry Identifier: KOFAM)
Record Dates: First submitted 2023-09-18; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Ventilation; Lung Function; Anesthesia, General
Keywords: Flow-controlled ventilation; High frequency jet ventilation; Lung protection; Laryngotracheal surgery
MeSH Terms: conditions — Respiratory Aspiration | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flow Controlled Ventilation Group (Experimental): Ventilation by Flow Controlled Ventilation mode Patient is scheduled for elective laryngotracheal surgery under general anesthesia. The ventilation mode for this group is Flow Controlled Ventilation mode.
  Interventions: Other: General anesthesia for laryngotracheal surgery; Other: Mechanical ventilation by FCV
- High Frequency Jet ventilation Group (Active Comparator): Ventilation by High Frequency Jet ventilation mode Patient is scheduled for elective laryngotracheal surgery under general anesthesia. The ventilation mode for this group is High Frequency Jet ventilation mode.
  Interventions: Other: General anesthesia for laryngotracheal surgery; Other: Mechanical ventilation by HFJV

INTERVENTIONS:
Other: General anesthesia for laryngotracheal surgery — Patients undergoing general anesthesia and mechanical ventilation.
Other: Mechanical ventilation by FCV — Mechanical ventilation is assured by Flow-controlled ventilation mode.
  Arms: Flow Controlled Ventilation Group
Other: Mechanical ventilation by HFJV — Mechanical ventilation is assured by High frequency jet ventilation mode.
  Arms: High Frequency Jet ventilation Group

SUMMARY:
Laryngotracheal surgery often requires a small diameter endotracheal tube to oxygenate patients under general anesthesia. Oxygenation is often only possible with high-frequency jet ventilators due to the use of small diameter and high resistance airway cannulas.

Flow controlled ventilation is a new ventilation modality capable for ventilation through a small diameter endotracheal tube (Tritube) with an active expiratory phase and the possibility of controlled carbon dioxide elimination during mechanical ventilation.

The aim of the present trial is to characterize perioperative changes in lung volume, ventilation inhomogeneity and respiratory mechanics in patients undergo upper airway surgery under general anesthesia with either flow controlled or high-frequency jet ventilation.

DETAILED DESCRIPTION:
This study is a randomized, controlled, assessor blind, monocentric study.

A new ventilation mode, called Flow Controlled Ventilation (FCV), has been suggested to minimize the amount of dissipated energy in the lungs and potentially could be protective during mechanical ventilation. FCV is unique in creating a stable gas flow into and also out of the patient's lungs to generate inspiration and expiration respectively. The FCV ventilation mode by its design allows the use of an ultrathin endotracheal tube with an inflatable cuff to secure the airways for ventilation. Therefore FCV offers several new surgical options for the treatment during laryngeal and tracheal surgery where the standard approach is usually the use of high-frequency jet ventilation (HFJV). The limitations of HFJV are however the lack of airway protection, limited monitoring of the respiratory variables and potential carbon dioxide (CO2) accumulation.

Participants for this study will be recruited at the University Hospitals of Geneva, scheduled for laryngotracheal surgery under general anesthesia. A total of 50 patients will be enrolled and randomly assigned into 2 groups: Group FCV (Flow controlled ventilation) and Group HFJV (high-frequency jet ventilation).

Measurements of functional residual capacity (FRC) and lung clearance index (LCI) will be performed in patients with a nitrogen multiple breath washout method, before and approximately 1 hour after surgery. Similarly, respiratory system resistance (R) and respiratory reactance (X) will be measured at the same time by using the Forced Oscillation Technique.

Relevance: There are no studies that addressed the value of flow controlled ventilation in terms of lung function parameters (FRC and LCI) and lung mechanics (R, X) in comparison to high-frequency jet ventilation in patients undergoing upper airway surgery.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed by the subject
* General anesthesia for laryngotracheal surgery
* Adult patients, female and male, over 18 years of age
* Elective surgery

Exclusion Criteria:

* Documented severe heart conditions (New York Heart Association Class 4, severe pulmonary hypertension)
* Documented severe respiratory disease (uncontrolled asthma, severe pulmonary fibrosis, chronic obstructive pulmonary disease GOLD 4)
* Documented severe Neurological diseases (Acute ischemic and hemorrhagic stroke within the preceding 3 months, uncontrolled seizures)
* Surgery that requires tracheotomy
* Obesity (Body Mass Index ≥ 30 kg/m2)
* Inability to follow the procedures of the study (mental condition or language barrier e.g. incomprehension of French language)
* Previous enrolment into the current study or other study that involves unknown medication in the past 12 months
* Allergy or contraindication to Propofol and/or Remifentanil and/or Rocuronium

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Alterations in the functional residual capacity (FRC) | Right before general anesthesia and approximately 1 hour after general anesthesia or before discharge from post anesthesia care unit
  FRC measured by the nitrogen multiple breath washout technique that will be applied before and after general anesthesia

SECONDARY OUTCOMES:
Alterations in the Lung clearance index (LCI) | Right before general anesthesia and approximately 1 hour after general anesthesia or before discharge from post anesthesia care unit
  LCI measured by the nitrogen multiple breath washout technique that will be applied before and after general anesthesia
Alterations in the respiratory resistance assessed by the forced oscillation technique (FOT) | Right before general anesthesia and approximately 1 hour after general anesthesia or before discharge from post anesthesia care unit
  Respiratory mechanics will be measured by the forced oscillation technique (FOT) to evaluate respiratory resistance (R).
Alterations in the respiratory reactance assessed by the forced oscillation technique (FOT) | Right before general anesthesia and approximately 1 hour after general anesthesia or before discharge from post anesthesia care unit
  Respiratory mechanics will be measured by the forced oscillation technique (FOT) to evaluate respiratory reactance (X).

OTHER OUTCOMES:
Changes in mean blood pressure | Intraoperative period with specific time points: before anesthesia induction, at the beginning of the surgery, at the end of surgery, right after extubation
  mean blood pressure (mmHg)
Changes in heart rate | Intraoperative period with specific time points: before anesthesia induction, at the beginning of the surgery, at the end of surgery, right after extubation
  heart rate (beat per minute)
Changes in oxygen saturation | Intraoperative period with specific time points: before anesthesia induction, at the beginning of the surgery, at the end of surgery, right after extubation
  Oxygen saturation will be measured by pulse oximetry (%)
Changes in transcutaneous carbon dioxide | Intraoperative period with specific time points: before anesthesia induction, at the beginning of the surgery, at the end of surgery, right after extubation
  Transcutaneous carbon dioxide will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Gergely Albu, MD, PhD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neder JA, Andreoni S, Castelo-Filho A, Nery LE. Reference values for lung function tests. I. Static volumes. Braz J Med Biol Res. 1999 Jun;32(6):703-17. doi: 10.1590/s0100-879x1999000600006. PMID 10412549
- [Background] Bourgain JL, Chollet M, Fischler M, Gueret G, Mayne A; membres du conseil du club en anesthesie en ORL. [Guide for the use of jet-ventilation during ENT and oral surgery]. Ann Fr Anesth Reanim. 2010 Oct;29(10):720-7. doi: 10.1016/j.annfar.2010.06.020. Epub 2010 Sep 15. French. PMID 20833503
- [Background] Bacher A, Pichler K, Aloy A. Supraglottic combined frequency jet ventilation versus subglottic monofrequent jet ventilation in patients undergoing microlaryngeal surgery. Anesth Analg. 2000 Feb;90(2):460-5. doi: 10.1097/00000539-200002000-00041. PMID 10648340
- [Background] Barnes T, van Asseldonk D, Enk D. Minimisation of dissipated energy in the airways during mechanical ventilation by using constant inspiratory and expiratory flows - Flow-controlled ventilation (FCV). Med Hypotheses. 2018 Dec;121:167-176. doi: 10.1016/j.mehy.2018.09.038. Epub 2018 Sep 24. PMID 30396474
- [Background] Tonetti T, Vasques F, Rapetti F, Maiolo G, Collino F, Romitti F, Camporota L, Cressoni M, Cadringher P, Quintel M, Gattinoni L. Driving pressure and mechanical power: new targets for VILI prevention. Ann Transl Med. 2017 Jul;5(14):286. doi: 10.21037/atm.2017.07.08. PMID 28828361
- [Background] Cressoni M, Gotti M, Chiurazzi C, Massari D, Algieri I, Amini M, Cammaroto A, Brioni M, Montaruli C, Nikolla K, Guanziroli M, Dondossola D, Gatti S, Valerio V, Vergani GL, Pugni P, Cadringher P, Gagliano N, Gattinoni L. Mechanical Power and Development of Ventilator-induced Lung Injury. Anesthesiology. 2016 May;124(5):1100-8. doi: 10.1097/ALN.0000000000001056. PMID 26872367
- [Background] Schmidt J, Wenzel C, Mahn M, Spassov S, Cristina Schmitz H, Borgmann S, Lin Z, Haberstroh J, Meckel S, Eiden S, Wirth S, Buerkle H, Schumann S. Improved lung recruitment and oxygenation during mandatory ventilation with a new expiratory ventilation assistance device: A controlled interventional trial in healthy pigs. Eur J Anaesthesiol. 2018 Oct;35(10):736-744. doi: 10.1097/EJA.0000000000000819. PMID 29734208
- [Background] Meulemans J, Jans A, Vermeulen K, Vandommele J, Delaere P, Vander Poorten V. Evone(R) Flow-Controlled Ventilation During Upper Airway Surgery: A Clinical Feasibility Study and Safety Assessment. Front Surg. 2020 Feb 28;7:6. doi: 10.3389/fsurg.2020.00006. eCollection 2020. PMID 32185179